CLINICAL TRIAL: NCT01601496
Title: Study of PERipheral Bypass GraFting: ProspECTive Evaluation of FUSION™ Vascular Graft for Above Knee Targets(PERFECTION)
Brief Title: Evaluation of FUSION™ Vascular Graft for Above Knee Targets
Acronym: PERFECTION
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow Enrollment
Sponsor: Maquet Cardiovascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VR7000856
Record Dates: First submitted 2012-04-23; First posted 2012-05-18 (Estimated); Results first posted 2020-10-14 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Peripheral Arterial Occlusive Disease (PAOD)
MeSH Terms: conditions — Peripheral Arterial Occlusive Disease 1

STUDY DESIGN:
Intervention Model Description: Patients treated with the FUSION Vascular Graft
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- FUSION Vascular Graft (Experimental): All subjects who received a FUSION Vascular Graft at the baseline implant procedure.
  Interventions: Device: FUSION Vascular Graft

INTERVENTIONS:
Device: FUSION Vascular Graft — All subjects who received the FUSION Vascular Graft at the baseline implant procedure.

SUMMARY:
The purpose of the post-market study was to evaluate the safety and performance of the FUSION Vascular Graft.

DETAILED DESCRIPTION:
This study was a prospective, single-arm, multicenter study conducted in Germany and Austria to evaluate the FUSION Vascular Graft in patients with peripheral arterial occlusive disease undergoing above-the-knee bypass. Follow-up visits were performed at 30 days, 6 months, 12 months and included patency and post operative complications not associated with bypass patency.

ELIGIBILITY:
Inclusion Criteria:

* No known malignant disease
* Patient was willing and able to have follow-up visits and examinations
* Peripheral arterial occlusive disease (PAOD) requiring treatment of the femoral artery; Fontaine stage IIb, III and IV with dry peripheral gangrene, and suitable for surgery
* Patient was not participating in other clinical trials that would conflict with this protocol
* Patient agreed to the study provisions and provided written informed consent

Exclusion Criteria:

* Urgent or emergent surgery of any kind
* Documented acute or suspected systemic infection
* Life expectancy of less than one year
* Patients who had a minor or major stroke within 6 weeks of the procedure or who had evidence of prior massive stroke
* Patients who had experienced a myocardial infarction within 6 weeks prior to the procedure or had unstable angina pectoris
* Severe chronic renal insufficiency or undergoing hemodialysis
* Patients treated with coumadin (warfarin) that had not been stopped within 72 before enrollment
* Medical conditions requiring oral anticoagulation
* Antiplatelet therapy with clopidogrel or dual antiplatelet as well as any other antithrombotic medication within 7 days prior to scheduled bypass surgery except unfractionated heparin or aspirin
* International normalized ratio (INR) > 2.0
* Known hypersensitivity to heparin
* Patient not tolerating aspirin
* Previous history of bypass surgery in the target limb
* Patient with category 6 ischemia (tissue loss)
* Acute limb ischemia of any grade (0-3)
* Patient with no outflow beyond the popliteal artery
* Pregnant or may become pregnant during the course of the study
* Uncontrolled arterial hypertension (BP > 200 mmHg) at 2 successive readings
* Anaemia (hemoglobin < 8 g/ml)
* Thrombocytopenia < 50 g/L
* Active bleeding according to clinical judgment
* Infected wet gangrene of any size and location at the target limb
* Compromised arterial flow
* Patient unwilling or unable to comply with follow-up requirements

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2009-10-26 (Actual); Primary Completion 2013-07-24 (Actual); Study Completion 2013-07-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Eckstein, Principal Investigator — Klinikum rechts der Isar; Afshin Assadian, MD, Principal Investigator — Wilhelminenspital Vienna
Locations (10):
- Wilhelminenspital Vienna, Vienna, Austria
- Germany (9):
  - Klinikum Darmstadt, Darmstadt
  - Universitätsklinikum Frankfurt, Frankfurt am Main
  - Klinikum Karlsruhe, Karlsruhe
  - Marienhospital Kevelaer, Kevelaer
  - Klinikum Ludwigsburg, Ludwigsburg
  - Klinikum München-Pasing, München
  - Klinikum rechts der Isar, München
  - Mathias-Spital, Rheine
  - Katharinenhospital, Stuttgart

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Assadian A, Eckstein HH; Peripheral Bypass Grafting: Prospective Evaluation of FUSION Vascular Graft for Above Knee Targets (PERFECTION) Study Group. Outcome of the FUSION vascular graft for above-knee femoropopliteal bypass. J Vasc Surg. 2015 Mar;61(3):713-9.e1. doi: 10.1016/j.jvs.2014.10.005. Epub 2014 Dec 10. PMID 25498193

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were referred to and treated at 10 vascular surgery centers in Germany and Austria. Enrolled subjects received a FUSION Vascular Graft between October 2009 and May 2012.
Pre-assignment Details: Patients were enrolled if they had peripheral artery occlusive disease (PAOD), signed informed consent forms, received subject numbers, and were screened for inclusion in the study. One subject failed to meet all eligibility criteria, prior to implantation of a FUSION vascular graft, and was not included in the efficacy or safety analyses.
Period: Overall Study
Arm/Group | FUSION Vascular Graft
Started | 117 (Enrolled)
Completed | 102 (Completed 12-M F/up)
Not Completed | 15
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 6
Not completed — Death | 4
Not completed — Other: patient refusal to continue | 3

BASELINE CHARACTERISTICS:
Population: Patients with peripheral vascular disease who underwent femoral-to-above-knee popliteal bypass with a FUSION Vascular Graft.
Arm/Group | FUSION Vascular Graft
Number analyzed (Participants) | 117
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.8 (8.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50
  Male | 67
Region of Enrollment [Number; unit: participants]
  Austria | 19
  Germany | 98
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 26.7 (4.36)
Ankle-brachial index [Mean (Standard Deviation); unit: ratio] — The Ankle-brachial index is the ratio between the systolic pressure measured at the ankle and the systolic pressure measured in the arm. Population: Patients with available measurement data for Ankle-brachial index.
  ratio
    number analyzed (Participants) | 115
    (all) | 0.53 (0.196)
Rutherford Category, No (%) [Count of Participants; unit: Participants] — Pre-Intervention Rutherford Classification Category, as assigned by Investigator. Higher grades represent more severe disease, ranging from asymptomatic (category 0) to major tissue loss (category 6).
  Participants
    Category 0, asymptomatic | 1
    Category 1, mild claudication | 1
    Category 2, moderate claudication | 55
    Category 3, severe claudication | 42
    Category 4, ischemic rest pain | 8
    Category 5, minor tissue loss | 10
    Category 6, major tissue loss | 0

OUTCOME MEASURES:

1. Primary Outcome: Participants With Primary Graft Patency at 12 Months
Description: Subjects were assessed to have had primary graft patency at 12 months. A graft was considered to have primary patency if it had remained continuously patent (i.e., had continued blood flow through it) from the time of implantation and it had uninterrupted patency with no interventions. Patency was assessed by duplex ultrasound imaging.
Time Frame: 12 Months
Population: Analysis limited to participants who were known primary patency failures (i.e. interventions were documented) or had a patency assessment at 12 months.
Measure: Count of Participants; unit: Participants
Arm/Group | FUSION Vascular Graft
Number analyzed (Participants) | 104
Participants | 89

2. Secondary Outcome: Participants With Secondary Graft Patency at 12 Months
Description: Subjects were assessed to have had secondary graft patency at 12 months. Secondary graft patency was defined as a graft patency established by another intervention to remediate occlusion within 12 months after surgery.
Time Frame: 12 Months
Population: Analysis limited to participants who had a patency assessment at 12 months or had been a secondary graft patency failure at a prior visit without restoration of flow.
Measure: Count of Participants; unit: Participants
Arm/Group | FUSION Vascular Graft
Number analyzed (Participants) | 103
Participants | 96

3. Secondary Outcome: Mean Ankle-brachial Index at 30 Days, 6 Months and 12 Months
Description: Ankle-brachial index at 30 days, 6 months, and 12 months. The ankle-brachial index is the ratio between the systolic pressure measured at the ankle and the systolic pressure measured in the arm.
Time Frame: 30 days, 6 months, 12 months
Population: Patients with available ankle-brachial index measurements at the individual time point. Note that the number of patients with an ankle-brachial index measurement varies by time point.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | FUSION Vascular Graft
Number analyzed (Participants) | 117
ratio
  30 days: number analyzed (Participants) | 104
  30 days | 0.97 (0.157)
  6 months: number analyzed (Participants) | 95
  6 months | 0.94 (0.210)
  12 Months: number analyzed (Participants) | 100
  12 Months | 0.91 (0.216)

4. Secondary Outcome: Rutherford Category at 30 Days, 6 Months and 12 Months
Description: Rutherford category at 30 days, 6 months and 12 months. Rutherford classification is a staging system to describe lower extremity ischemia, and is assigned by the Investigator. Higher grades represent more severe disease, ranging from asymptomatic (category 0) to major tissue loss (category 6).
Time Frame: 30 days, 6 months, 12 months
Population: Patients with available Rutherford classification at the individual time point. Note that the number of patients with an assigned Rutherford classification varies by time point.
Measure: Count of Participants; unit: Participants
Arm/Group | FUSION Vascular Graft
Number analyzed (Participants) | 117
Participants
  30 Days: number analyzed (Participants) | 107
  30 Days: Category 0, asymptomatic | 65
  30 Days: Category 1, mild claudication | 30
  30 Days: Category 2, moderate claudication | 8
  30 Days: Category 3, severe claudication | 3
  30 Days: Category 4, ischemic rest paint | 0
  30 Days: Category 5, minor tissue loss | 1
  30 Days: Category 6, major tissue loss | 0
  6 Months: number analyzed (Participants) | 97
  6 Months: Category 0, asymptomatic | 67
  6 Months: Category 1, mild claudication | 23
  6 Months: Category 2, moderate claudication | 3
  6 Months: Category 3, severe claudication | 1
  6 Months: Category 4, ischemic rest paint | 1
  6 Months: Category 5, minor tissue loss | 2
  6 Months: Category 6, major tissue loss | 0
  12 Months: number analyzed (Participants) | 102
  12 Months: Category 0, asymptomatic | 68
  12 Months: Category 1, mild claudication | 20
  12 Months: Category 2, moderate claudication | 7
  12 Months: Category 3, severe claudication | 3
  12 Months: Category 4, ischemic rest paint | 3
  12 Months: Category 5, minor tissue loss | 1
  12 Months: Category 6, major tissue loss | 0

5. Secondary Outcome: Number of Participants Experiencing Major Adverse Limb Events and Periprocedural Death
Description: Major Adverse Limb Events (MALE) were defined as major amputation (any amputation that resulted in limb shortening) or major graft reintervention (including placement of a new bypass graft at the same anatomic site, a jump/interposition graft, graft thrombectomy, graft excision (explant), or graft thrombolysis). Periprocedural Death (POD) was defined as death within 30 days of the index procedure or within 30 days of any remedial procedure performed at the same anatomical site or as a result of the initial procedure.
Time Frame: 12 Months
Population: All subjects who received a FUSION Vascular Graft at the baseline implant procedure.
Measure: Count of Participants; unit: Participants
Arm/Group | FUSION Vascular Graft
Number analyzed (Participants) | 117
Participants
  Major amputation | 0
  Procedure-related death | 0
  Major graft reintervention | 15
  Any MALE or POD | 15

ADVERSE EVENTS:
Time Frame: Through 12 months follow up
Groups:
- FUSION Vascular Graft: All subjects who receive a FUSION Vascular Graft at the baseline implant procedure
Arm/Group | FUSION Vascular Graft
All-Cause Mortality (participants affected / at risk) | 4/117
Serious Adverse Events (participants affected / at risk) | 48/117
Other Adverse Events (participants affected / at risk) | 0/117
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FUSION Vascular Graft (N=117)
Cardiac Failure (Cardiac disorders) | 1 (2)
Gallstone ileus (Gastrointestinal disorders) | 1 (1)
Ileal stenosis (Gastrointestinal disorders) | 2 (3)
Death (General disorders) | 1 (1)
Impaired healing (General disorders) | 2 (2)
Oedema peripheral (General disorders) | 2 (2)
Renal failure (Renal and urinary disorders) | 1 (1)
Graft infection (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Wound infection (Infections and infestations) | 8 (8)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 3 (3)
Transplant failure (Injury, poisoning and procedural complications) | 1 (1)
Vascular graft occlusion (Injury, poisoning and procedural complications) | 15 (24)
Wound secretion (Injury, poisoning and procedural complications) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Angioplasty (Surgical and medical procedures) | 1 (1)
Aortic aneurysm repair (Surgical and medical procedures) | 1 (1)
Peripheral endarterectomy (Surgical and medical procedures) | 1 (1)
Surgery (Surgical and medical procedures) | 1 (1)
Aortic stenosis (Vascular disorders) | 2 (3)
Intermittent claudication (Vascular disorders) | 1 (1)
Haematoma (Vascular disorders) | 4 (4)
Leriche syndrome (Vascular disorders) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1)
Peripheral ischemia (Vascular disorders) | 2 (2)
Vasculitis (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No